CLINICAL TRIAL: NCT02789059
Title: Muscle Oxygenation Modification During Effort in 4 Groups of Neuromuscular Diseases Compared to Healthy Controls, and Mitochondrial Function and Phenotype Assessment
Brief Title: Muscle Oxygenation in Effort in Neuromuscular Diseases
Acronym: OXYNEMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013_29; 2014-A01157-40 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Diseases
Keywords: Becker muscular dystrophy; Facioscapulohumeral dystrophy; congenital myopathy; motor neurone diseases
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Dystrophy, Duchenne; Myotonia Congenita; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- muscle oxygenation (Experimental): assesment of muscle oxygenation and gas exchanges
  Interventions: Other: muscle oxygenation

INTERVENTIONS:
Other: muscle oxygenation — Subjects will be invited to perform an isokinetic effort of the knee extensors against an isokinetic dynamometer. During this effort, muscle oxygenation and oxygen consumption will be assessed with a near infrared spectroscopy device and a gas exchange measurement device. Patients affected by Becker muscular dystrophy and healthy controls will be invited to have a muscle biopsy of the vastus lateralis.
  Other Names: Muscle biopsy

SUMMARY:
Previous studies showed modifications of muscle oxygenation parameters in muscular dystrophies du to an impairment or an absence of dystrophin.

Our study aim at assessing muscle oxygenation during effort in different neuromuscular diseases (muscular dystrophies related and not related to dystrophin, non dystrophic myopathies and motor neuron diseases) compared to a group of healthy controls. Patients and controls are invited to perform an inframaximal , standardized effort of the knee extensors by the mean of an isokinetic dynamometer. Muscle oxygenation parameters are assessed through a Near Infrared Spectroscopy (NIRS) Device.

In patients affected by dystrophin related myopathies, a muscle biopsy will be performed in order to analyse mitochondrial oxygenation parameters and mitochondrial phenotype.

Our Hypothesis is that muscle oxygenation is impaired in dystrophin related muscular dystrophies compared to other neuromuscular diseases and healthy controls because of lack of muscle capillary vessels dilatation during effort and impairment of mitochondrial function.

DETAILED DESCRIPTION:
This study is a prospective physiological study in a pathological condition (neuromuscular diseases).

5 groups of voluntary participants will be investigated:

1. 20 subjects affected by Dystrophin related muscular dystrophy (Becker Muscular Dystrophy ) 2. Subjects affected by muscular dystrophy not related to dystrophin impairment : 20 subjects affected by facioscapulohumeral dystrophy and 20 subjects affected by Limb Girdle Muscular dystrophy 3. 20 subjects affected by non-dystrophic myopathies (Congenital myopathies ) 4. 20 subjects affected by motor diseases: amyotrophic lateral sclerosis(ALS), Charcot Marie Tooth disease, Spinal Muscular Atrophy .

5. 20 healthy controls Objective: asses the muscular oxygenation modifications during a standardized effort and compare the variables between groups. Analyze the mitochondrial function and phenotype in the BMD group compared to healthy controls Outcome : Muscle Oxygenation by Near Infrared Spectroscopy parameters; oxygen consumption, Muscle Function Measure, Vignos and Brooke score, Borg scale, 6 minutes walk test, mitochondrial phenotype, mitochondrial oxygenation 3 visits : 1- inclusion 2- standardized effort protocol 3- for Becker dystrophy patients and voluntary controls, muscle biopsy of the Vastus Lateralis

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects and
* subjects affected by one of the fallowing neuromuscular diseases: Becker Muscular dystrophy Facioscapulohumeral dystrophy, Limb Girdle Muscular Dystrophy , Congenital Myopathy , Spinal Muscular Atrophy Charcot Marie Tooth Disease and Amyotrophic Lateral Sclerosis ,
* able to walk
* presenting a manual muscle testing of at Least 4/5 on the quadriceps according to the Medical research Council

Exclusion Criteria:

* musculoskeletal pain of the quadriceps
* other neurological disorders
* Heart failure arrhythmia, uncontrolled hypertension, angina pectoris
* dyspnoea >2 according to the NYHA
* Peripheral artery disease
* BMI >30kg.m-2.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
muscle oxygenation | on the day of first evaluation Visit V1
  level of deoxyhemoglobin assessed with the NIRS device during the isokinetic effort of the knee extensors
Muscle oxygenation | on the day of first evaluation Visit V1
  kinetics of the deoxyhemoglobin assessed with the NIRS device during the isokinetic effort of the knee extensors

SECONDARY OUTCOMES:
maximal isokinetic strength of the knee extensors | on the day of first evaluation Visit V1
  measurements of the maximal moment during a maximal effort of the knee extensors with an isokinetic dynamometer
Gas exchange | on the day of first evaluation Visit V1
  measurements of O2 and CO2 exchanges during the isokinetic effort
MFM score | on the day of first evaluation Visit V1
  Motor Function Measure score (in %) assessment. quantitative scale that makes it possible to measure the functional motor abilities of a person affected by a neuromuscular disease.
6 Minutes Walking Test (MWT) | on the day of first evaluation Visit V1
  assessment of the time performed during a 6 minutes walking test
Vignos functional scales | on the day of first evaluation Visit V1
  assesment of the 1 to 6 Vignos score for the lower limb functional assesment
Brooke functional scales | on the day of first evaluation Visit V1
  the 1 to 10 Brooke score for upper limb functional assesment
Medical Research Council Muscle testing | on the day of first evaluation Visit V1
  Assesment of the Medical Research Council 1 to 5 Muscle testing score of the quadriceps muscles
Mitochondrial phenotype | at V2 at least 1 week after V1
  Mitochondrial respiration (O2 consumption) of muscle fibers of the vastus lateralis
Mitochondrial H2O2 production | at V2 at least 1 week after V1
  Mitochondrial H2O2 production of muscle fibers of the vastus lateralis
kinetic of Muscle oxygenation | on the day of first evaluation Visit V1
  kinetic of level of deoxyhemoglobin during the isokinetic effort of the extensors of the knee

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Tiffreau, MD, Principal Investigator — CHRU de LILLE
Locations (3):
- France (3):
  - Hôpital Amiens Nord, Service de Neurologie, Amiens
  - CHRU de Lille, Hôpital Swyngedhauw, Lille
  - Hôpital Sébastopol, CHU de Reims, Reims

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allart E, Olivier N, Hovart H, Thevenon A, Tiffreau V. Evaluation of muscle oxygenation by near-infrared spectroscopy in patients with Becker muscular dystrophy. Neuromuscul Disord. 2012 Aug;22(8):720-7. doi: 10.1016/j.nmd.2012.04.011. Epub 2012 Jun 8. PMID 22683375